CLINICAL TRIAL: NCT04169815
Title: Pivotal Evaluation of the Access Natriuretic Peptdie Assay(s) as an Aid in the Diagnosis and Assessment of Severity of Acute Heart Failure - Emergency Department Subject Enrollment and Specimen Collection
Brief Title: Access Natriuretic Peptide Assay(s) Pivotal - Emergency Department Subject Enrollment and Specimen Collection
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HF-01-19
Record Dates: First submitted 2019-11-17; First posted 2019-11-20 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
Keywords: Natriuretic Peptide
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and Plasma sample collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- ED Setting: An acute HF population enrolled at the emergency department. Testing of clinical samples will be performed with the Access natriuretic peptide assay.
  Interventions: Diagnostic Test: Access Immunodiagnostic Products

INTERVENTIONS:
Diagnostic Test: Access Immunodiagnostic Products — Access Natriuretic Peptide Assay

SUMMARY:
The purpose of the pivotal study is to collect blood specimens and clinical data from patients suspected of having Heart Failure (HF), which will be tested at a future date on Natriuretic Peptide assay(s) to validate diagnostic cutoffs and assess HF severity.

DETAILED DESCRIPTION:
A prospective clinical sample collection and future natriuretic peptide testing will be conducted in an emergency department only population. Patients presenting to the Emergency Department (ED) with signs and symptoms of acute heart failure will be approached for enrollment.

Clinical and laboratory data will be collected to establish product performance and clinical concordance to adjudicated clinical diagnosis. Approximately 1800 evaluable subjects at geographically dispersed sites in the US will be enrolled in the study.

Sample collection and testing of clinical samples with the Access Natriuretic Peptide assay will be performed under two separate protocols

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained
* Adult aged 21 years or older
* Presenting with a clinical suspicion of acute HF
* Subject clinical history available for review by Sponsor or delegates and FDA or other regulatory agencies

Exclusion Criteria:

* Dyspnea clearly not secondary to HF (e.g. primary lung disease or chest trauma)
* Stage 4 or 5 Chronic Kidney Disease (CKD)
* Chronic dialysis
* Participation in a clinical study that may interfere with participation in this study
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be representative of an acute heart failure population enrolled at Emergency Departments. Patients presenting with a suspicion of acute heart failure will be approached for enrollment.
Sampling Method: Probability Sample
Enrollment: 2370 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the future Natriuretic Peptide Assay(s) | Single blood draw upon study entry at day 1
  Establish the performance of the future Natriuretic Peptide assay(s) against the adjudicated diagnosis.

SECONDARY OUTCOMES:
Heart Failure Severity Assessment | Single blood draw upon study entry at day 1 and two remote follow up visits
  Demonstrate that the Access Natriuretic Peptide Assay may be used for assessment of heart failure severity.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Beckman Coulter Site AJ, Loma Linda, California
  - Beckman Coulter Site AL, Sacramento, California
  - Beckman Coulter Site AB, Gainesville, Florida
  - Beckman Coulter Site AG, Indianapolis, Indiana
  - Beckman Coulter Site AN, Kansas City, Kansas
  - Beckman Coulter Site AA, Detroit, Michigan
  - Beckman Coulter Site AH, St Louis, Missouri
  - Beckman Coulter Site AI, Albuquerque, New Mexico
  - Beckman Coulter Site AE, Stony Brook, New York
  - Beckman Coulter Site AK, Cleveland, Ohio
  - Beckman Coulter Site AF, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Beckman Coulter Site AC, Charleston, South Carolina
  - Beckman Coulter Site AD, Nashville, Tennessee
  - Beckman Coulter Site AM, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iwanaga Y, Nishi I, Furuichi S, Noguchi T, Sase K, Kihara Y, Goto Y, Nonogi H. B-type natriuretic peptide strongly reflects diastolic wall stress in patients with chronic heart failure: comparison between systolic and diastolic heart failure. J Am Coll Cardiol. 2006 Feb 21;47(4):742-8. doi: 10.1016/j.jacc.2005.11.030. Epub 2006 Jan 26. PMID 16487838
- [Background] Kinnunen P, Vuolteenaho O, Ruskoaho H. Mechanisms of atrial and brain natriuretic peptide release from rat ventricular myocardium: effect of stretching. Endocrinology. 1993 May;132(5):1961-70. doi: 10.1210/endo.132.5.8477647.
- [Background] Mueller T, Gegenhuber A, Poelz W, Haltmayer M. Diagnostic accuracy of B type natriuretic peptide and amino terminal proBNP in the emergency diagnosis of heart failure. Heart. 2005 May;91(5):606-12. doi: 10.1136/hrt.2004.037762. PMID 15831643
- [Background] Friedewald VE Jr, Burnett JC Jr, Januzzi JL Jr, Roberts WC, Yancy CW. The editor's roundtable: B-type natriuretic peptide. Am J Cardiol. 2008 Jun 15;101(12):1733-40. doi: 10.1016/j.amjcard.2008.03.017. Epub 2008 Apr 22. No abstract available. PMID 18549849
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Januzzi JL, van Kimmenade R, Lainchbury J, Bayes-Genis A, Ordonez-Llanos J, Santalo-Bel M, Pinto YM, Richards M. NT-proBNP testing for diagnosis and short-term prognosis in acute destabilized heart failure: an international pooled analysis of 1256 patients: the International Collaborative of NT-proBNP Study. Eur Heart J. 2006 Feb;27(3):330-7. doi: 10.1093/eurheartj/ehi631. Epub 2005 Nov 17. PMID 16293638
- [Background] Maisel AS, Krishnaswamy P, Nowak RM, McCord J, Hollander JE, Duc P, Omland T, Storrow AB, Abraham WT, Wu AH, Clopton P, Steg PG, Westheim A, Knudsen CW, Perez A, Kazanegra R, Herrmann HC, McCullough PA; Breathing Not Properly Multinational Study Investigators. Rapid measurement of B-type natriuretic peptide in the emergency diagnosis of heart failure. N Engl J Med. 2002 Jul 18;347(3):161-7. doi: 10.1056/NEJMoa020233. PMID 12124404